CLINICAL TRIAL: NCT05089279
Title: An Open Label, Randomized, Single-dose, 2-sequence, 2-period, Cross-over Phase 1 Study to Evaluate the Safety and Pharmacokinetics of CKD-349 in Healthy Adult Volunteers
Brief Title: Study to Evaluate the Safety and Pharmacokinetics of CKD-349 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A111_01BE2019
Record Dates: First submitted 2021-10-14; First posted 2021-10-22 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2021-12

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): Period 1: D113/ Period 2: CKD-349
  Interventions: Drug: D113; Drug: CKD-349
- Sequence2 (Experimental): Period 1: CKD-349/ Period 2: D113
  Interventions: Drug: D113; Drug: CKD-349

INTERVENTIONS:
Drug: D113 — QD, PO
Drug: CKD-349 — QD, PO

SUMMARY:
Study to Evaluate the Safety and Pharmacokinetics of CKD-349

DETAILED DESCRIPTION:
An Open Label, Randomized, Single-dose, 2-sequence, 2-period, Cross-over Phase 1 Study to Evaluate the Safety and Pharmacokinetics of CKD-349 in Healthy Adult Volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers aged ≥ 19 years
2. Weight ≥50kg (man) or 45kg (woman), with calculated body mass index (BMI) of 18 to 30 kg/m2
3. Those who have no congenital diseases or chronic diseases and have no abnormal symptoms or findings.
4. Those who are eligible for clinical trials based on laboratory (hematology, blood chemistry, serology, urology) and 12-lead ECG results at screening.
5. Those who agree to contraception until 7 days after clinical trial.
6. Individuals who voluntarily decide to participate and agree to comply with the cautions after fully understand the detailed description of this clinical trial.

Exclusion Criteria:

1. Those who have clinically significant diseases or history in digestive systems, cardiovascular system, endocrine system, respiratory system, blood·tumor, infectious disease, kidney and urogenital system, mental·nervous system, musculoskeletal system, immune system, otolaryngology, skin system, ophthalmology system, etc.
2. Those who have a history of gastrointestinal surgery except simple appendectomy and hernia surgery.
3. Those who take barbiturate and any related drugs which may cause induction or inhibition of drug metabolism within 1 month before the first administration of investigational products or take drugs that may interfere with this clinical trials within 10 day before the first administration
4. Those who received investigational products or participated in bioequivalence tests within 6 months before the first administration of clinical trial drugs.
5. Those who donated whole blood within 8 weeks or donated ingredients within 2 weeks, or received a blood transfusion within 4 weeks.
6. Those who exceed an alcohol and cigarette consumption than below criteria A. Alcohol: Man- 21 glasses/week, Woman - 14 glasses/week (1 glass: Soju 50mL, Wine 30mL, or beer 250mL) B. Smoking: 20 cigarettes/day
7. Those who overreacts to the ingredient of this drug and is administering an angiotensin conversion enzyme (ACE) inhibitor or has not passed 36 hours since discontinuation of administration and has a history of vascular edema when administering an angiotensin conversion enzyme (ACE) inhibitor or an angiotensin receptor antagonist (ARB).
8. Those who are deemed insufficient to participate in this clinical study by investigators.
9. Woman who are pregnant or breastfeeding.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-04-06 (Actual)

PRIMARY OUTCOMES:
AUCt of CKD-349 | 0, 0.08, 0.17, 0.33, 0.5, 0.67, 0.83, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 48 hours
  AUCt: Area under the concentration-time curve from time zero to time
Cmax of CKD-349 | 0, 0.08, 0.17, 0.33, 0.5, 0.67, 0.83, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 48 hours
  Cmax: Maximum plasma concentration of the drug

SECONDARY OUTCOMES:
AUCinf of CKD-349 | 0, 0.08, 0.17, 0.33, 0.5, 0.67, 0.83, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 48 hours
  Area under the concentration-time curve from zero up to ∞
Tmax of CKD-349 | 0, 0.08, 0.17, 0.33, 0.5, 0.67, 0.83, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 48 hours
  Time to maximum plasma concentration
AUCt/AUCinf of CKD-349 | 0, 0.08, 0.17, 0.33, 0.5, 0.67, 0.83, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 48 hours
  AUCt/AUCinf
T1/2 of CKD-349 | 0, 0.08, 0.17, 0.33, 0.5, 0.67, 0.83, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 48 hours
  Terminal elimination half-life

CONTACTS AND LOCATIONS:
Overall Officials: JaeWoo Kim, Principal Investigator — Study Principal Investigator
Locations (1):
- H Plus Yangji Hospital, Seoul, Gwanak-gu, South Korea